CLINICAL TRIAL: NCT05800938
Title: The Effect of Oral Isosorbide Mononitrate Therapy on Umbilical Artery Doppler Resistance Index in Pregnancies With Intrauterine Growth Restriction: Prospective Randomized Control Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, MayaAbdElRazek, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS 382/ 2022
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isosorbid mononitrate group (Active Comparator): Imdur 30 mg tablet AstraZeneca egypt twice daily for 4 weeks
  Interventions: Drug: Isosorbid mononitrate
- placebo group (Placebo Comparator): Tablets twice daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isosorbid mononitrate — Imdur tablets were given twice daily for 4 weeks
  Other Names: Isosorbide -5- mononitrate biphasic; Imdur
  Arms: Isosorbid mononitrate group
Drug: Placebo — Placebo tablets were given twice daily for 4 weeks
  Arms: placebo group

SUMMARY:
Will follow up umblical artery Doppler indices for pregnancies with iugr taking placebo and oral isosorbide mononitrate to study its efficacy on the intrauterine growth restricted fetuses

DETAILED DESCRIPTION:
Patients meeting these criteria are to be randomized into one of the following two groups:

* Group A (n=23): The Isosorbide Mononitrate group: will receive (IMDUR®, 30 mg, tablet, AstraZeneca, Egypt) (Isosorbide-5-mononitrate Biphasic) twice daily for 4-6 weeks (according to xPharm: The Comprehensive Pharmacology Reference, 2007, Pages 1-4).
* Group B (n=23): The placebo group will receive (Osteocare®, tab, VITABIOTICS, Egypt) twice daily for 4-6 weeks Justification: Using PASS 11 program for sample size calculation, setting power at 80% and alpha error at 0.05 and according to "Trapani et al., 2015", the expected change in UTA-PI in isosorbide mononitrate group=21% compared to no change in placebo group. Sample size of 23 women per group will be needed to detect difference between two groups.

The study is to be double-blinded, where neither the researcher, nor the participants will know what type of medication each participant will receive, as a nurse will give each patient a closed envelope containing 21 tablets of one of the above two medications in a randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

* age : 18-34 BMI: 18-30 Singleton pregnancy Gestational age between 28-30 Criteria of IUGR

Exclusion Criteria:

Had known or suspected chromosomal or structural anomaly Had a condition which will require delivery Multiple pregnancy

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Reduction in umbilical artery Doppler indices | 4 weeks after initiation of treatment
  Measuring of the umbilical artery Doppler resistant index (RI) with the patient in semi recombinant position, during a period of absent fetal movement and breathing. a minimum of three uniform Doppler waveforms will be measured

SECONDARY OUTCOMES:
Enhancement of fetal growth as measured by the increase in estimated fetal weight and abdominal circumference | 4 weeks after initiation of treatment
  Estimation of fetal weight calculated automatic in the software of the ultrasound scanner utilizing Hadlock's formula (Biparital diameter BPD, Femur length FL, Abdominal circumference AC).
Development of fetal complications | 4 weeks after initiation of treatment
  IUFD, Fetal distress or deterioration of Doppler indices requiring delivery
Interval to delivery | 37 weeks
  gestational age at delivery in weeks
Maternal side effects | 4 weeks after initiation of treatment
  Headache, palpitation, postural hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt